CLINICAL TRIAL: NCT02350348
Title: NECTARINE: NEonate-Children sTudy of Anaesthesia pRactice IN Europe Epidemiology of Morbidity and Mortality in Neonatal Anaesthesia: A European Prospective Multicentre Observational Study
Brief Title: NEonate-Children sTudy of Anaesthesia pRactice IN Europe Epidemiology of Morbidity and Mortality in Neonatal Anaesthesia
Acronym: NECTARINE
Status: Completed | Type: Observational
Sponsor: European Society of Anaesthesiology (Other)
Responsible Party: Sponsor
Other Study IDs: NECTARINE
Record Dates: First submitted 2015-01-15; First posted 2015-01-29 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2020-07

CONDITIONS: Children; Anaesthesia
Keywords: neonates; infants; anaesthesia; mortality; adverse effects; Epidemiological Study; European Society of Anaesthesiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To study the 30-day morbidity and mortality after neonatal anaesthesia, and predictive factors that can be responsible for poor outcome.

DETAILED DESCRIPTION:
The recent pharmacological and technological advancements are making paediatric anaesthesia safer, minimizing thereby the risk of serious adverse events. Despite recent advancements, there is still a significant incidence of life-threatening complications following general and regional anaesthesia without complete identification of predictive factors. Several cohort studies reported the incidence of perioperative anaesthetic complications, but the results were generally limited to a single centre.

Hence, a prospective multicentre study "APRICOT" has been recently conducted in order to establish the incidence of some severe critical events and to identify the risk factors for their occurrence [ClinicalTrials.gov identifier # NCT01878760]. This European Society of Anaesthesiology Clinical Trial Network project is currently in progress with over 300 participating centres and more than 25,000 patients, from birth to 15 years of age, to be included. The NECTARINE is specifically focussed on the neonatal population.

The NECTARINE aims to include all neonates and infants from birth to 60 weeks of postmenstrual age scheduled for an elective or urgent diagnostic or surgical procedure under sedation or general anaesthesia with or without regional analgesia or under regional anaesthesia. The primary aim of this study is to identify the occurrence of peri-anaesthesia (during and up to the first 120 minutes) interventions needed to treat or improve one of the following: (1) airway management, (2) oxygenation, (3) alveolar ventilation, (4) glycaemia and Na+, (5) cardiovascular instability, (6) body temperature, (7) brain oxygenation, and (8) anaemia. The parameter or the clinical event that has triggered the intervention will be specifically reported. As secondary aims the in- and out- of hospital morbidity and mortality will be studied at 30 and 90 days from anaesthesia.

Following sample size estimation, the plan is to recruit between 5000 children over a period of twelve consecutive weeks, including weekends and after-hours across the 30 European countries represented at the European Society of Anaesthesiology Council or part of geographical Europe.

The 12-week recruitment period will be chosen by each site commencing on 1 January 2016.The last possible inclusion date will be decided by the Study Steering Committee depending on the recruitment rate. Participating hospitals will be provided with data acquisition sheets that enable anonymous standardized recording of all patients' parameters, which will be used by the local institution to fill in the electronic case report form.

Descriptive statistical analysis will be performed for the primary endpoint (occurrence of severe critical events and 95% confidence interval). Univariate and multivariate analysis will be performed to test factors associated with the endpoint. Results of logistic regression will be reported as adjusted odds ratio (OR) with 95 % confidence intervals .

ELIGIBILITY:
Inclusion Criteria:

* children from birth to 60 weeks of post-menstrual age undergoing anaesthesia for surgical or diagnostic procedures admitted to participating centres during a predetermined 12-week recruitment period
* all elective inpatient or outpatient surgical procedures performed under general anaesthesia with or without regional analgesia, or under regional anaesthesia alone;
* all diagnostic procedures performed under general anaesthesia;
* all urgent or emergency procedures performed in- or out-of-hours.
* all procedures performed in Neonatal Intensive Care Unit (NICU) / Paediatric Intensive Care Unit (PICU) or directly admitted from intensive care to the operating room

Exclusion Criteria:

- Infants aged over 60 weeks of age on the day of surgery.

Max Age: 60 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates and infants from birth to 60 weeks of post-menstrual age
Sampling Method: Non-Probability Sample
Enrollment: 5500 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
The incidence of interventions performed by the anaesthesia team in response to (i) a critical event or (ii) a major change of physiological parameters during anaesthesia management. | Anaesthesia time : up to 120 minutes post-anaesthesia either in Post Anesthesia Care Unit (PACU) or neonatal ward
  This is a composite that will include several physiological parameters to be observed: (1) airway management, (2) oxygenation, (3) alveolar ventilation, (4) glycaemia and Na+, (5) cardiovascular instability, (6) body temperature, (7) brain oxygenation, and (8) anaemia.

SECONDARY OUTCOMES:
The incidence of adverse events | 120 minutes post-anaesthesia either in Post Anesthesia Care Unit (PACU) or neonatal ward
  This is a composite that will include:
  * Unplanned delayed extubation.
  * Need for ECMO (extracorporeal membrane oxygenation).
  * Need for chest left open (for cardiac surgery only).
  * Unplanned hospital admission (originally scheduled as outpatient)
Mortality | up to 30 days after anaesthesia
  As determined from medical records
Morbidity | at 30 days after anaesthesia
  as determined from medical records: until discharge or at 30 days if still in hospital.
In- and out-hospital mortality | 90 days after anaesthesia
  As determined from medical records
In- and out-hospital morbidity | 90 days after anaesthesia
  As determined from medical records

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Disma, MD, Study Chair — Dept. Anesthesia - Istituto G. Gaslini - Genoa - Italy
Locations (10):
- Cliniques Universitaires St Luc, Brussels, Belgium
- Odense University Hospital, Odense, Denmark
- Cnopf'sche Kinderklinik/Klinik Hallerwiese, Nuremberg, Germany
- Instituto Giannina Gaslini, Genoa, Italy
- Wilhelmina Childrens Hospital, Utrecht, Netherlands
- Clinical University Hospital Department of Anaesthesiology and Intensive Care, Wroclaw, Poland
- University Childrens hospital, Belgrade, Serbia
- Geneva University Hospitals, Geneva, Switzerland
- United Kingdom (2):
  - Royal Aberdeen Children's Hospital, Aberdeen
  - Great Ormond St Hospital for Children's NHS, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Disma N, Leva B, Dowell J, Veyckemans F, Habre W. Assessing anaesthesia practice in the vulnerable age group: NECTARINE: A European prospective multicentre observational study. Eur J Anaesthesiol. 2016 Apr;33(4):233-5. doi: 10.1097/EJA.0000000000000414. No abstract available. PMID 26928166
- [Derived] Neumann C, Schenk A, Schindler E, Becke-Jakob K; German Nectarine Group Collaborators. Epidemiology, Morbidity and Mortality Associated With Anesthesia in Early Life: A Subgroup Analysis of the German NEonate and Children audiT of Anesthesia pRactice IN Europe (NECTARINE) Cohort. Paediatr Anaesth. 2026 Jan 16. doi: 10.1002/pan.70115. Online ahead of print. PMID 41546183
- [Derived] Fuchs A, Disma N, Engelhardt T, Marchesini V, Riedel T, Boda K, Habre W, Riva T; NECTARINE Steering Committee; NECTARINE Group of the European Society of Anaesthesiology and Intensive Care Clinical Trial Network. Ventilation strategies and risk factors for intraoperative respiratory critical events and postoperative pulmonary complications in neonates and small infants: a secondary analysis of the NECTARINE cohort☆. Br J Anaesth. 2025 Nov;135(5):1528-1536. doi: 10.1016/j.bja.2024.12.038. Epub 2025 Feb 20. PMID 39979152
- [Derived] Disma N, Engelhardt T, Hansen TG, de Graaff JC, Virag K, Habre W; NECTARINE Group of the European Society of Anaesthesiology and Intensive; AUSTRIA (Maria Vittinghoff); BELGIUM (Francis Veyckemans); CROATIA (Sandra Kralik); CZECH REPUBLIC (Jiri Zurek); DENMARK (Tom Hansen); ESTONIA (Reet Kikas); FINLAND (Tuula Manner); FRANCE (Christophe Dadure, Anne Lafargue); GERMANY (Karin Becke, Claudia Hoehne); GREECE (Anna Malisiova); HUNGARY (Andrea Szekely); IRELAND (Brendan O'Hare); ITALY (Nicola Disma); LATVIA (Zane Straume); LITHUANIA (Laura Lukosiene); LUXEMBOURG (Bernd Schmitz); MALTA (Francis Borg); NETHERLANDS (Jurgen de Graaff); NORWAY (Wenche B Boerke); POLAND (Marzena Zielinska); PORTUGAL (Maria Domingas Patuleia); ROMANIA (Radu Tabacaru); SERBIA (Dusica Simic); SLOVAKIA (Miloslav Hanula); SLOVENIA (Jelena Berger); SPAIN (Ignacio Galvez Escalera); SWEDEN (Albert Castellheim); SWITZERLAND (Walid Habre); TURKEY (Dilek Ozcengiz - Zehra Hatipoglu); UKRAINE (Dmytro Dmytriiev); UNITED KINGDOM (Thomas Engelhardt, Suellen Walker); Management Team. Neonates undergoing pyloric stenosis repair are at increased risk of difficult airway management: secondary analysis of the NEonate and Children audiT of Anaesthesia pRactice IN Europe. Br J Anaesth. 2022 Nov;129(5):734-739. doi: 10.1016/j.bja.2022.07.041. Epub 2022 Sep 6. PMID 36085092
- [Derived] Fuchs A, Disma N, Virag K, Ulmer F, Habre W, de Graaff JC, Riva T; NECTARINE Group of the European Society of Anaesthesiology and Intensive Care Clinical Trial Network. Peri-operative red blood cell transfusion in neonates and infants: NEonate and Children audiT of Anaesthesia pRactice IN Europe: A prospective European multicentre observational study. Eur J Anaesthesiol. 2022 Mar 1;39(3):252-260. doi: 10.1097/EJA.0000000000001646. PMID 34845167
- [Derived] Disma N, Veyckemans F, Virag K, Hansen TG, Becke K, Harlet P, Vutskits L, Walker SM, de Graaff JC, Zielinska M, Simic D, Engelhardt T, Habre W; NECTARINE Group of the European Society of Anaesthesiology Clinical Trial Network; Austria; Belgium; Croatia; Czech Republic; Denmark; Estonia; Finland; France; Germany; Greece; Hungary; Ireland; Italy; Latvia; Lithuania; Luxembourg; Malta; Netherlands; Norway; Poland; Portugal; Romania; Serbia; Slovakia; Slovenia; Spain; Switzerland; Turkey; Ukraine; United Kingdom. Morbidity and mortality after anaesthesia in early life: results of the European prospective multicentre observational study, neonate and children audit of anaesthesia practice in Europe (NECTARINE). Br J Anaesth. 2021 Jun;126(6):1157-1172. doi: 10.1016/j.bja.2021.02.016. Epub 2021 Apr 1. PMID 33812668
- [Derived] Disma N, Virag K, Riva T, Kaufmann J, Engelhardt T, Habre W; NECTARINE Group of the European Society of Anaesthesiology Clinical Trial Network; AUSTRIA (Maria Vittinghoff); BELGIUM (Francis Veyckemans); CROATIA (Sandra Kralik); CZECH REPUBLIC (Jiri Zurek); DENMARK (Tom Hansen); ESTONIA (Reet Kikas); FINLAND (Tuula Manner); FRANCE (Christophe Dadure, Anne Lafargue); GERMANY (Karin Becke, Claudia Hoehne); GREECE (Anna Malisiova); HUNGARY (Andrea Szekely); IRELAND (Brendan O'Hare); ITALY (Nicola Disma); LATVIA (Zane Straume); LITHUANIA (Laura Lukosiene); LUXEMBOURG (Bernd Schmitz); MALTA (Francis Borg); NETHERLANDS (Jurgen de Graaff); NORWAY (Wenche B Boerke); POLAND (Marzena Zielinska); PORTUGAL (Maria Domingas Patuleia); ROMANIA (Radu Tabacaru); SERBIA (Dusica Simic); SLOVAKIA (Miloslav Hanula); SLOVENIA (Jelena Berger); SPAIN (Ignacio Galvez Escalera); SWEDEN (Albert Castellheim); SWITZERLAND (Walid Habre); TURKEY (Dilek Ozcengiz - Zehra Hatipoglu); UKRAINE (Dmytro Dmytriiev); UNITED KINGDOM (Thomas Engelhardt, Suellen Walker); Management Team. Difficult tracheal intubation in neonates and infants. NEonate and Children audiT of Anaesthesia pRactice IN Europe (NECTARINE): a prospective European multicentre observational study. Br J Anaesth. 2021 Jun;126(6):1173-1181. doi: 10.1016/j.bja.2021.02.021. Epub 2021 Apr 1. PMID 33812665